CLINICAL TRIAL: NCT00447993
Title: A Phase II/III Study of Encapsulated Human NTC-201 Cell Implants Releasing Ciliary Neurotrophic Factor (CNTF) for Participants With Retinitis Pigmentosa Using Visual Acuity as the Primary Outcome
Brief Title: A Study of Encapsulated Cell Technology (ECT) Implant for Patients With Late Stage Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNTF 3
Record Dates: First submitted 2007-03-09; First posted 2007-03-15 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; eye disease; retinal disorder; CNTF
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases; Retinal Diseases | interventions — Ciliary Neurotrophic Factor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Low Dose NT-501 (Experimental): NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
  Interventions: Combination Product: Low Dose NT-501
- High Dose NT-501 (Experimental): NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
  Interventions: Combination Product: High Dose NT-501

INTERVENTIONS:
Combination Product: Low Dose NT-501 — Low Dose NT-501 Implanted in study eye and fellow eye received sham surgery
  Other Names: CNTF implant
  Arms: Low Dose NT-501
Combination Product: High Dose NT-501 — High Dose NT-501 Implanted in study eye and fellow eye received sham surgery
  Other Names: CNTF implant
  Arms: High Dose NT-501

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of CNTF implants on vision in persons with retinitis pigmentosa, Usher type II & III, and Choroideremia. This research is being done because there are no effective therapies for people with these retinal degenerations. They are genetic disorders that affect our ability to see at night, and later cause tunnel vision and loss of central vision. Retinal degenerations affect the retina, a light sensitive layer of cells in the back of the eye. Slowly over time, these cells die and cause permanent loss of vision.

The implant is a small capsule that contains human retinal pigment epithelium cells. These cells have been given the ability to make CNTF and release it through the capsule membrane into the surrounding fluid. This study will look at the effect of the implant on vision loss by retinitis pigmentosa, Usher type II & III, and Choroideremia. In this study, two different CNTF dose levels will be used: a high dose and a low dose in one eye, as well as a sham (or placebo) surgery in the other eye.

DETAILED DESCRIPTION:
This study will involve about 16 visits over 1½ years for specific tests of the participant's vision and health. These visits may include visual exams, blood draw for laboratory testing, brief medical history and exam, and occasionally a questionnaire (survey), in addition to the visit for the surgical procedures. The primary effectiveness outcome for this study will be a visual acuity score one year after the implant surgery. There will be about 13 centers participating in this study, and up to 60 people enrolled across the US. Each participant joining the study who has completed initial screening will then be scheduled to have a brief surgical procedure performed on each eye, one of which will include a very small cell-filled implant. Follow-up visits for repeat assessments will be required regularly to determine if the implant being tested is safe and effective for use to treat RP.

ELIGIBILITY:
Inclusion Criteria:

1. Participant was older than 18, but less than 68 years of age.
2. Participant understood and signed the informed consent. If the participant's vision was impaired to the point where he/she could not read the informed consent document, the document would be read to the participant in its entirety.
3. Females of childbearing potential (women with last menses <1 year prior to screening) agreed to use an effective form of birth control from study onset until they completed the 18-month study visit.
4. Participant was medically able to undergo ophthalmic surgery for the NT-501 device.
5. Participant's clinical diagnosis was consistent with retinal degeneration in the set of retinitis pigmentosa (RP) dystrophies characterized by the following features:

   1. clinical evidence of progressive photoreceptor cell dysfunction and degeneration of the outer retina.
   2. intraretinal bone-spicule'-like pigment observed in clinical examination (not necessarily applicable to choroideremia).
   3. peripheral visual field constriction documented on standard testing.
   4. symptomatic night blindness.
   5. reduction of both rod and cone electroretinogram (ERG) responses. Individuals diagnosed with Retinitis Pigmentosa, Usher Syndrome Type 2 or Type 3 (without profound deafness or cochlear implant) or with Choroideremia (CHM) and who met the inclusion criteria were considered as potential candidates for this study. A maximum of 5 Usher Syndrome Type 2 or Type 3 and a maximum of 5 Choroideremia participants could be enrolled in this trial.
6. Each eye had a visual acuity score of at least 24 (20/320) and no more than 63 (20/63) letters.
7. Each eye had an ERG amplitude reduced below the 95% limit of normal (CI) per site by Full Field 28-32 Hz flicker.

Exclusion Criteria:

1. Participant was medically unable to comply with study procedures or follow-up visits.
2. Participant had glaucoma (defined as independent optic atrophy causing vision loss), irrespective of whether it was currently treated or untreated.
3. Participant had classic syndromic RP.
4. Participant had optic nerve atrophy beyond modest pallor, primary cone-rod dystrophy, unilateral bulls-eye maculopathy, cystoid maculopathy as judged by OCT reading center, or other retinal dystrophy.
5. Participant who had any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 3, or a nuclear opacity > standard 3 as measured on the AREDS clinical lens grading system.
6. Participant had chronic requirement (e.g., > or =4 weeks at a time) for ocular medications or has disease(s) that in the judgment of the examining physician were vision threatening, toxic to the lens, retina, or optic nerve or might affect the primary outcome.
7. Participant had a requirement of acyclovir and/or related products during study duration.

   To be eligible for this study, the participant must have discontinued use of these products prior to enrollment and must not continue with the products until after they had completed the study.
8. Participant had evidence of corneal opacification or lack of optical clarity.
9. Participant had undergone lens removal in the last 3 months, with or without intra-ocular lens implantation, or had undergone intra-ocular lens replacement within 6 months prior to enrollment.
10. Participant was receiving systemic steroids or other immunosuppressive medications.
11. Participant had undergone LASIK surgery or other refractive surgery for either eye in less than 6 months prior to screening.
12. Participant was currently participating in or had participated in any other clinical trial of a drug by ocular or systemic administration within the last 6 months.
13. Participant had previous exposure to an intra-ocular device or implant into the eye (excluding intra-ocular lens).
14. Participant had uveitis or other retinal inflammatory disease.
15. Participant was receiving oral or other insulin treatment for diabetes.
16. Participant who had a history of myocardial infarction within the last 12 months.
17. Participant was pregnant or lactating.
18. Participant was considered immunodeficient or had a known history of HIV. A laboratory test for HIV was performed, and a positive result was also an exclusion criterion.
19. Participant with a history of ocular herpes zoster.
20. Participant was on chemotherapy.
21. Participant had a history of malignancy, except study participants having cancer treated successfully ≥5 years prior to inclusion in the trial.
22. Participant with severe hearing disabilities in both ears.
23. Participant with diabetic retinopathy in either eye.
24. Participant had history of retinal detachment in either eye.
25. Participant had been diagnosed and treated for amblyopia as an infant.
26. Participant with a history of Pars Plana Vitrectomy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-01-08 (Actual); Primary Completion 2009-05-26 (Actual); Study Completion 2009-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Birch, MD, Principal Investigator — Retina Foundation of the Southwest
Locations (11):
- United States (11):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of Califoria, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Retina Group of Florida, Hollywood, Florida
  - University of Florida, Jacksonville, Florida
  - Kellogg Eye Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - NY University Medical Center, New York, New York
  - Casey Eye Institue, Portland, Oregon
  - The Hamilton Eye Institute, Memphis, Tennessee
  - Retina Foundation of Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birch DG, Weleber RG, Duncan JL, Jaffe GJ, Tao W; Ciliary Neurotrophic Factor Retinitis Pigmentosa Study Groups. Randomized trial of ciliary neurotrophic factor delivered by encapsulated cell intraocular implants for retinitis pigmentosa. Am J Ophthalmol. 2013 Aug;156(2):283-292.e1. doi: 10.1016/j.ajo.2013.03.021. Epub 2013 May 10. PMID 23668681
- [Derived] Kauper K, McGovern C, Sherman S, Heatherton P, Rapoza R, Stabila P, Dean B, Lee A, Borges S, Bouchard B, Tao W. Two-year intraocular delivery of ciliary neurotrophic factor by encapsulated cell technology implants in patients with chronic retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7484-91. doi: 10.1167/iovs.12-9970. PMID 23049090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total number of participant in the low dose group was 22 and the high dose group was 45 since each patient consented to treatment in one eye and sham treatment in the other eye.
Units Other Than Participants: Eyes
Groups:
- Low Dose Arm - Implant: NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- Low Dose Arm - Sham: Sham Implant in Fellow Eye (Low Dose Arm)
- High Dose Arm - Implant: NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- High Dose Arm - Sham: Sham Implant in Fellow Eye (High Dose Arm)
Period: Overall Study
Arm/Group | Low Dose Arm - Implant | Low Dose Arm - Sham | High Dose Arm - Implant | High Dose Arm - Sham
Started | 22; 22 Eyes | 22; 22 Eyes | 45; 45 Eyes | 45; 45 Eyes
Completed | 22; 22 Eyes | 22; 22 Eyes | 41; 41 Eyes | 41; 41 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 4; 4 Eyes | 4; 4 Eyes
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Total number of participants in the trial was 67, with 22 participants in the Low Dose Arm and 45 participants in the High Dose Arm. Note, the participants also received a sham surgery in fellow eye on both study arms, which was used as reference therapy. No capsule was implanted in fellow eye. Baseline reports include sham as a separate column for each arm.
Units Other Than Participants: Eyes
Groups:
- High Dose: NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- Total: Total of all reporting groups
Arm/Group | Low Dose Arm - Implant | Low Dose Arm - Sham | High Dose | High Dose Arm - Sham | Total
Number analyzed (Participants) | 22 | 22 | 45 | 45 | 67
Number analyzed (Eyes) | 22 | 22 | 45 | 45 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (10.5) | 41.1 (10.5) | 42.0 (11.0) | 42.0 (11.0) | 41.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 25 | 25 | 66
  Male | 14 | 14 | 20 | 20 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 2 | 10
  Not Hispanic or Latino | 19 | 19 | 43 | 43 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 2 | 2 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 4 | 10
  White | 18 | 18 | 39 | 39 | 114
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ocular History - Years Since RP Diagnosis [Mean (Standard Deviation); unit: Years] | 24.66 (9.55) | 24.66 (9.55) | 21.50 (13.21) | 21.50 (13.21) | 22.52 (12.17)
Type of Ocular History [Count of Units; unit: Eyes]
  Ocular Disease | 22 | 22 | 45 | 45 | 134
  Ocular Surgery | 11 | 9 | 21 | 21 | 62
  Ocular Treatment | 2 | 2 | 2 | 2 | 8
BCVA Letter Score [Mean (Standard Deviation); unit: Letters] — BCVA = best corrected visual acuity; For BCVA, baseline=average of values at Baseline Visits 2 and 3 Population: Two patients, both in the high dose were randomized but did not receive the implant and did not take part in the study. One of these participants ended study participation prior to completion of Visit 3 baseline visit. The other patient is included in the BCVA baseline data set; however, did not proceed with surgery.
  Letters
    number analyzed (Participants) | 22 | 22 | 44 | 44 | 66
    number analyzed (Eyes) | 22 | 22 | 44 | 44 | 132
    (all) | 45.5 (11.2) | 44.8 (10.4) | 45.0 (10.4) | 46.7 (9.1) | 45.5 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Change in Best-corrected Visual Acuity (BCVA) Using the Electronic Visual Acuity (EVA) Technology at Month 12.
Description: The primary efficacy endpoint was the proportion of patients demonstrating an improvement in best-corrected visual acuity (BCVA), defined as an increase of 10 letters or more at the 1-Year post-implant visit (pre-explant, if explant is completed). No response is defined as an improvement of <10 letters.
Time Frame: 12 months post-implant
Population: Results are based on participants who completed the 1-yr post implant visit/assessment.
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Low Dose Arm - Implant | Low Dose Arm - Sham | High Dose | High Dose Arm - Sham
Number analyzed (Participants) | 21 | 21 | 42 | 42
Number analyzed (Eyes) | 21 | 21 | 42 | 42
participants
  Response (Greater than or equal to 10 letter improvement) | 1 | 1 | 3 | 1
  No Response | 20 | 20 | 39 | 41

2. Secondary Outcome: Number of Participants With and Without Best Corrected Visual Acuity Response Over the 18-month Follow-up Period (Months 1, 3, 6, 12 and 18)
Description: The key visits for efficacy assessments were Months 1, 3, 6, 12 and 18. At these time points, BCVA was measured 3 times and the mean outcome reported. The assessments were conducted by masked technicians. The change from baseline for BCVA was summarized by time. Response is defined as an improvement in visual acuity by an increase of 10 letters or more whereas no response is <10 letters.
Time Frame: From initial implant to 18 months post-implant
Population: Data set provides details for each timepoint based on number of patients who completed BCVA procedure at the each applicable visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Arm - Implant | Low Dose Arm - Sham | High Dose | High Dose Arm - Sham
Number analyzed (Participants) | 22 | 22 | 43 | 43
Participants
  1 month post-implant: Response | 1 | 1 | 3 | 1
  1 month post-implant: No Response | 21 | 21 | 40 | 42
  3 months post-implant: Response: number analyzed (Participants) | 22 | 22 | 42 | 42
  3 months post-implant: Response | 2 | 1 | 2 | 0
  3 months post-implant: No Response: number analyzed (Participants) | 22 | 22 | 42 | 42
  3 months post-implant: No Response | 20 | 21 | 40 | 42
  6 months post-implant: Response: number analyzed (Participants) | 21 | 21 | 42 | 42
  6 months post-implant: Response | 1 | 0 | 4 | 2
  6 months post-implant: No Response: number analyzed (Participants) | 21 | 21 | 42 | 42
  6 months post-implant: No Response | 20 | 21 | 38 | 40
  12 months post-implant: Response: number analyzed (Participants) | 21 | 21 | 42 | 42
  12 months post-implant: Response | 1 | 1 | 3 | 1
  12 months post-implant: No Response: number analyzed (Participants) | 21 | 21 | 42 | 42
  12 months post-implant: No Response | 20 | 20 | 39 | 41
  18 months post-implant: Response: number analyzed (Participants) | 19 | 19 | 32 | 32
  18 months post-implant: Response | 0 | 2 | 2 | 0
  18 months post-implant: No Response: number analyzed (Participants) | 19 | 19 | 32 | 32
  18 months post-implant: No Response | 19 | 17 | 30 | 32

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of the consent through 18 months post-implant.
Groups:
- Low Dose: NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
- High Dose: NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=22) | High Dose (N=22)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=22) | High Dose (N=43)
Abnormal sensation in eye (Eye disorders) | 2 (2) | 2 (2)
Anterior chamber cell (Eye disorders) | 7 (7) | 12 (12)
Anterior chamber flare (Eye disorders) | 5 (5) | 10 (10)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Conjunctival cyst (Eye disorders) | 2 (2) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 16 (16) | 32 (32)
Conjunctival Hyperaemia (Eye disorders) | 11 (11) | 15 (15)
Conjunctival Oedema (Eye disorders) | 2 (2) | 6 (6)
Eye inflammation (Eye disorders) | 2 (2) | 4 (4)
Eye irritation (Eye disorders) | 1 (1) | 3 (3)
Eye pain (Eye disorders) | 2 (2) | 7 (7)
Eye pruritis (Eye disorders) | 1 (1) | 4 (4)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 10 (10)
Macular Oedema (Eye disorders) | 0 (0) | 3 (3)
Maculopathy (Eye disorders) | 2 (2) | 1 (1)
Miosis (Eye disorders) | 1 (1) | 11 (11)
Pupils unequal (Eye disorders) | 2 (2) | 5 (5)
Vision blurred (Eye disorders) | 3 (3) | 3 (3)
Visual acuity reduced (Eye disorders) | 0 (0) | 3 (3)
Vitreous detachment (Eye disorders) | 0 (0) | 3 (3)
Vitreous disorder (Eye disorders) | 3 (3) | 7 (7)
Vitreous opacities (Eye disorders) | 1 (1) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Suture related complication (Injury, poisoning and procedural complications) | 10 (10) | 11 (11)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes